CLINICAL TRIAL: NCT01941017
Title: Evaluation of the Ovarian Reserve in Infertile Patients With Endometriosis
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, karim H abdel-maeboud, Professor, Ain Shams University
Other Study IDs: EORIE
Record Dates: First submitted 2013-03-27; First posted 2013-09-13 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2013-09

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Minimal or mild endometriosis: Patients with minimal or mild endometriosis diagnosed via laparoscopy.
- Tubal obstruction without endometriosis: Patients with tubal obstruction due to infection or adhesion with absent evidence for endometriosis on laparoscopy

SUMMARY:
Comparison between Ovarian reserve markers in patients with minimal/mild endometriosis and patients with tubal factor infertility

DETAILED DESCRIPTION:
Comparison between Ovarian reserve markers (laboratory or us) in patients with minimal/mild endometriosis and patients with tubal factor infertility including:

Cycle Day 2 or 3 FSH and E2, Serum AMH and antral follicular count

ELIGIBILITY:
Inclusion Criteria:

Age 18-35 years of age. Written and signed informed consent by the patient to participate in the study. Patients with regular menses, both ovaries, serum TSH within normal range, body mass index (BMI) <30 kg/m2 with normal sperm analysis of the husband.

Exclusion Criteria:

Patients with previous endocrine disorders. Cases in which the cause for infertility was other than endometriosis (except for patients with tubal obstruction, in the control group).

Patient with previous surgery for endometriosis.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Group I : patients with minimal or mild endometriosis (I or II) as proven by laparoscopy (n=20).
  Group II: (control group) patients with tubal obstruction without endometriosis (n=20).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2009-04; Primary Completion 2011-11 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Assessment of ovarian reserve in the 2 groups | 2 years
  Serum AMH and antral follicular count (AFC)

SECONDARY OUTCOMES:
Other Hormonal parameters | 2 years
  Cycle day 2 or 3 FSH and E2